CLINICAL TRIAL: NCT04153916
Title: Artificial Eye Blinking Stimulation Following Paralysis of the Facial Nerve
Acronym: Bioniceye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurotrigger Ltd (Industry)
Collaborators: Tel Aviv Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0266-19-TLV
Record Dates: First submitted 2019-10-27; First posted 2019-11-06 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2021-09

CONDITIONS: Facial Paralysis; Bell Palsy
Keywords: Eye blinking, facial nerve paralysis, nano electrode
MeSH Terms: conditions — Facial Paralysis; Bell Palsy

STUDY DESIGN:
Intervention Model Description: elicit a complete or a partial eyelid closure & To optimize the location of the Neurotrigger's electrodes, and define the level of the pain generated, if any, during device implementation and stimulation, as well as the method for the personal adjustment of the precise pattern of stimulation (strength, intensity, other features) to achieve eye blinking for different patients.
Masking Description: The Principle Investigators of the Clinical study will code the patients by the study enrolment number provided at the day of enrolment and is not disclosed to the sponsor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single use and continuous use (Other): Patients with a continuous unilateral facial paralysis that underwent an operation for facial reanimation will be enrolled at least one year after the operation according to review of medical records of the Department of plastic surgery.
  Patients with temporary unilateral facial paralysis secondary to Bell's palsy as was identified in the admission to the Hospital Department of Plastic Surgery or to the Department of Ear, Nose and Throat.
  Interventions: Device: Neurotrigger eye blinking stimulator

INTERVENTIONS:
Device: Neurotrigger eye blinking stimulator — Phase 1 - The first stage is composed of a one-time participation for about three hours and involves:
  1. Verifying compliance of the patients with the research inclusion and exclusion criteria
  2. Completion of the study clinical report form (CRF) for this stage
  3. Placement of the single use mini-electrodes that will be adhered to the facial skin near the non-blinking eye and coupled to the Neurotrigger stimulator to elicit eyelid closure.
  Participants may be enrolled to the second phase up to one year from the first phase visit In the second stage the duration of the participation is about three weeks (six days a week) and includes daily use of the device for up to 10 hours a day. During nights the patient will continue is standard pattern of either eye closure or leaving the eye open, as the patient used to do prior to the study.
  This stage will involve a patient with a partner that is designated to support the patient closely during the placement and adjustment of the system

SUMMARY:
Artificial eye blinking stimulation following damage to the facial nerve. Group 1 - Patients with a persistent unilateral facial paralysis (palsy) that underwent an operation for facial reanimation Group 2 - Patients with temporary unilateral facial paralysis, secondary to unilateral Bell's palsy.

Primary objective: To evaluate whether the Neurotigger device can elicit a complete or a partial eyelid closure of the affected eye.

Secondary objective: To optimize the location of the Neurotrigger's electrodes, and define the level of the pain generated, if any, during device implementation and stimulation, as well as the method for the personal adjustment of the precise pattern of stimulation (strength, intensity, other features) to achieve eye blinking for different patients.

DETAILED DESCRIPTION:
The study will involve two groups:

Group 1: Patients with a continuous unilateral facial paralysis that underwent an operation for facial reanimation will be enrolled at least one year after the operation according to review of medical records of the Department of plastic surgery.

Group 2: Patients with temporary unilateral facial paralysis secondary to Bell's palsy as was identified in the admission to the Hospital Department of Plastic Surgery or to the Department of Ear, Nose and Throat.

After being identified eligible to participate in the study, the patients will be invited to join the study, sign on the written informed consent, and their demographic and medical history will be recorded.

Patients identified to belong to these study groups in other hospitals may join the study, after pre-evaluation and medical record analysis by the study Principle Investigator (PI)/Co-PI.

The study will be constructed in two phases:

Phase 1 - The first stage is composed of a one-time participation for about three hours. This feasibility stage involves:

1. Verifying compliance of the patients with the research inclusion and exclusion criteria
2. Completion of the study clinical report form (CRF) for this stage
3. Placement of the single use mini-electrodes that will be adhered to the facial skin near the non-blinking eye and coupled to the Neurotrigger stimulator to elicit eyelid closure.

An initial report will then be issued to summarize the patient's experience of using the system in the first testing attempt to identify a complete or partial eye blinking.

Participants identified to respond to the stimulator at a partial or complete eye closure level, will be invited to continue to use the device for additional two hours in the hospital premises.

A summary meeting will then be held to issue a summary report covering the overall patient's experience of using the system throughout the testing period.

The purpose of this first stage is to examine the possibility of closing the patient eyelid completely or partially, optimize electrode position, and maximize the patient's comfort level.

A profile of system efficacy in generating eyelid closure will then be generated including the characterization of the stimulus pattern (intensity, frequency, etc.)

Phase 2: The purpose of this stage is to examine how a continued use of the device by the patient may improve outcomes, and reduce complications that are derived of the facial nerve paralysis

Participants may be enrolled to the second phase up to one year from the first phase visit

In this second stage the duration of the participation is about three weeks (six days a week) and includes daily use of the device for up to 10 hours a day. During nights the patient will continue is standard pattern of either eye closure or leaving the eye open, as the patient used to do prior to the study.

This stage will involve a patient with a partner that is designated to support the patient closely during the placement and adjustment of the system.

The patient and the partner will both obtain a detailed mutual training of placing the electrode and device, activating the device (partner) and its use (patient) to assure complete assistance and guidance in installing the system and its use.

Prior to starting this stage the patient will undergo eye examination and will complete a Patient Graded Instrument for Facial Nerve Paralysis - The FaCE Scale Questionnaire - to evaluate the life quality with the facial nerve paralysis (Laryngoscope. 2001 Mar;111(3):387-98.Validation of a patient-graded instrument for facial nerve paralysis: the FaCE scale. Kahn JB et al.)

Patients are provided with help desk number to answer questions and queries during the study period as needed.

They will get a clear guidance of the possibility to get support at home by experience system user or by phone-call or by videoconference (Skype or the like) by communicating with the experienced Sponsor's personnel who can help them adjust the electrode to the face and reducing discomfort.

In case of a skin rush or any skin discomfort, the patient will call the clinic and will be invited to medical examination and, if necessary, for treatment of a rush reducing and calming ointment and be advised of re-using the system.

Participants will make an intermediate evaluation at one and a half week and a final visit at three weeks.

The last visit will include eye examination to compare the eye functioning before and after Phase 2, and the completion of a FaCE Scale Questionnaire to evaluate potential improvement in life quality.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet ALL of the following criteria will be eligible for enrollment into this study:

All patients

1. Male or female above 18 years of age inclusive
2. All patients will have to agree to provide a written informed consent, Fully understand all elements of and actually sign and date the written Institutional Review Board (IRB) approved informed consent before initiation of protocol-specified procedures;
3. Willing to provide medical and demographic records of their facial paralysis, the consequences of the paralysis and general medical history.

Group 1:

5. Patients who comply with the definition of continuous existing unilateral facial paralysis and who underwent an operation for facial reanimation at least one year prior to enrollment

Group 2:

5. Patients who comply with the definition of temporary unilateral facial paralysis secondary to Bell's palsy up to 2 years from the event.

Second Phase

1. All initial inclusion criteria will be as in phase 1
2. Enrollment will be dependent on having a partner willing and capable to offer the six days a week daily support in placing the Neurotrigger simulator and closing eye at night time for a period of 3 weeks.

Exclusion Criteria:

1. Patients with chronic facial paralysis and secondary established damage to the eye occurring prior to enrollment, Who did not undergo facial reanimation surgery.
2. Patients with psychiatric, addictive, or any other disorder that compromises ability to give genuine informed consent for participation in this study.
3. Patients suffering from any skin condition that will prevent effective attachment of the electrodes, including but not limited to allergy to any of the components of the skin electrode.
4. Woman who is pregnant (positive pregnancy test)
5. Woman who is nursing
6. Unwillingness or inability to follow the procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Eyelid closure - Partial or complete closure | 3 hours
  Partial or complete eye closure. The results will be detailed in a data table which will include details of the number of participants, affiliation to a research group and level of eyelid closure.

SECONDARY OUTCOMES:
Stage 2 only - Improving quality of life - The measurement will be performed by filling out a Quality of Life Questionnaire. | three weeks
  Reducing dry eye effects. Dry eye effects will be measured by filling out a Quality of Life Questionnaire including questioning about the frequency of use of eye drops.

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Gur, MD, Principal Investigator — Chairman, Dep. Plastic Surgery, Tel Aviv Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center (Ichilov), Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
The product is protected by PCT application number: PCT/IL2019/050819 Study results will be published in medical journals

REFERENCES:
- Available data/document: Study Protocol: 0266-19-TLV — http://www.neurotrigger.info — Upon completion of the study, results will be published and the study data will be available from the PI